CLINICAL TRIAL: NCT00773838
Title: An International, Multicenter, Open-Label Study of Vorinostat (MK0683) in Combination With Bortezomib in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Vorinostat (MK0683), an Histone Deacetylase (HDAC) Inhibitor in Combination With Bortezomib in Patients With Relapsed or Refractory Multiple Myeloma (MK-0683-095)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-095; 2008-003753-33 (EudraCT Number); MK-0683-095 (Other: Merck); 2008_524 (Other: Merck)
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Vorinostat; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat + Bortezomib (Experimental): Participants receive vorinostat 400 mg, orally, once daily (QD) on Days 1-14 of each 21-day treatment cycle and bortezomib 1.3mg/m^2 intravenous (IV) injection QD on Days 1, 4, 8 and 11 of each 21-day treatment cycle for up to 26 cycles. Participants with progressive disease (PD) after 2 cycles of treatment or no change (NC) after 4 cycles of treatment receive additional treatment of Dexamethasone, 20 mg of total daily dose, orally on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day treatment cycle for up to 26 cycles. Eligible participants could receive additional treatment on an extension.
  Interventions: Drug: Vorinostat; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Vorinostat — Four 100 mg vorinostat capsules orally, once daily (QD) by mouth on Days 1-14 of each 21-day treatment cycle.
  Other Names: MK-0683; Suberoylanilide hydroxamic acid; Zolinza
Drug: Bortezomib — Bortezomib 1.3 mg/m^2, IV injection QD on Days 1, 4, 8, and 11 of each 21-day treatment cycle.
  Other Names: Velcade
Drug: Dexamethasone — Five 4 mg Dexamethasone tablets orally, QD on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day treatment cycle if PD is observed after 2 treatment cycles or if NC to disease is observed after 4 treatment cycles.
  Other Names: Decadron

SUMMARY:
The purpose of this study is to evaluate the clinical activity of vorinostat in combination with bortezomib in participants with relapsed or refractory multiple myeloma after at least 2 prior treatment regimens. The primary objective is to define the objective response rate (RR) associated with the administration of vorinostat in combination with bortezomib to patients with relapsed and refractory multiple myeloma after at least 2 prior treatment regimens. The primary hypothesis of the study is the administration of vorinostat in combination with bortezomib will result in a clinically meaningful rate of objective response.

DETAILED DESCRIPTION:
The protocol has been amended to indicate that the Final Analysis is designated as the time when the primary endpoint of 29 responders has been met, or the time when all participants have discontinued treatment or have been enrolled in the study for at least 6 months (if the primary endpoint is not reached by this time). Following the Final Analysis, participants will be allowed to continue study treatment in an extension as long as they have not met the criteria for discontinuation, and will be followed for overall survival and serious AEs.

ELIGIBILITY:
Inclusion Criteria:

* Has an established diagnosis of multiple myeloma based on myeloma diagnostic criteria
* Must have adequate organ function
* Is refractory to prior bortezomib regimen and have also been exposed to prior Immunomodulatory imide drugs (IMiD: thalidimide or lenalidmide)
* Has relapsed and refractory multiple myeloma after at least 2 prior treatment regimens
* Has performance status of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Has measurable disease, defined as any quantifiable serum monoclonal (M) protein value and, where applicable, urine light chain of ≥200 mg/24 hours
* Female participants are not pregnant and not breastfeeding, and are not a woman of childbearing potential (WOCBP) or are a WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 30 days after the last dose of study intervention
* Male participants must agree to use approved contraception during the treatment period and for at least 30 days after the last dose of study intervention and refrain from donating sperm during this period
* Is relapsed, refractory, intolerant, and/or ineligible (in the opinion of the investigator) to other therapies including an IMiD (thalidomide or lenalidomide)
* Is refractory to bortezomib (no response on prior bortezomib containing regimen or progression on or within 60 days of bortezomib containing regimen

Exclusion Criteria:

* Has known hypersensitivity to any components of bortezomib or vorinostat
* Has had a prior allogeneic bone marrow transplant or plans to undergo any type of bone marrow transplantation within 4 weeks of the initiation of study therapy
* Has an active systemic infection
* Has acute diffuse infiltrative pulmonary disease or pericardial disease
* Has known hypersensitivity to any components of bortezomib or vorinostat
* Has active Hepatitis B or C, plasma cell leukemia, or is human immunodeficiency virus (HIV) positive
* Has history of a prior malignancy with the exception of cervical intraepithelial neoplasia; non-melanoma skin cancer; adequately treated localized prostate carcinoma with prostate specific antigen (PSA) < 0.1; or who has undergone potentially curative therapy with no evidence of that disease for five years, or who is deemed at low risk for recurrence by his/her treating physician
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has plasma cell leukemia defined as the presence of more than 20% plasma cells in the peripheral blood and an absolute plasma cell count of at least 2000/μL
* Has a history of a gastrointestinal surgery or other procedures that might, in the opinion of the Investigator, interfere with the absorption or swallowing of the study drug
* Has preexisting National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Grade 1 neuropathy with pain or >Grade 2 neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2011-05-16 (Actual); Study Completion 2012-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Siegel DS, Dimopoulos M, Jagannath S, Goldschmidt H, Durrant S, Kaufman JL, Leleu X, Nagler A, Offner F, Graef T, Eid JE, Houp J, Gause C, Vuocolo S, Anderson KC. VANTAGE 095: An International, Multicenter, Open-Label Study of Vorinostat (MK-0683) in Combination With Bortezomib in Patients With Relapsed and Refractory Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2016 Jun;16(6):329-334.e1. doi: 10.1016/j.clml.2016.02.042. Epub 2016 Mar 4. PMID 27025160

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 143 participants enrolled, 142 participants were allocated to treatment. Five participants received additional treatment for about 1 year during an extension as per investigator's discretion based on clinical benefit of the treatment received. All 5 participants discontinued extension treatment and were followed for survival up to 2 years post last dose of treatment.
Period: Overall Study
Arm/Group | Vorinostat + Bortezomib
Started | 143
Completed | 0
Not Completed | 143
Not completed — Adverse Event | 29
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 8
Not completed — Progressive Disease | 82
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 21

BASELINE CHARACTERISTICS:
Population: All allocated participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 143
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 138
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 34
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 102
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (RR)
Description: Objective RR was defined as percentage (%) of participants with complete response (CR: disappearance of original monoclonal (M) paraprotein from blood & urine on at least 2 determinations for at least 6 weeks (WKs) by immunofixation studies, <5% plasma cells in bone marrow on at least 1 determination, no increase in size/number of lytic bone lesions (LBLs) & disappearance of soft tissue plasmacytomas (STP) for at least 6 WKs on skeletal survey (SS) if available) or partial response (PR: ≥50% reduction in serum M protein for at least 2 determinations 6 WKs apart, if present, reduction in 24-hour urinary light chain excretion by ≥90% or ≤200 mg for at least 2 determinations 6 WKs apart, ≥50% reduction in STP size for at least 6 WKs, & no increase in size/number of LBLs on SS if available) as assessed by Independent Adjudication Committee (IAC) per European Blood & Marrow Transplant (EBMT) criteria. To report RR & 95% confidence intervals (CIs), exact test of binomial parameter was used.
Time Frame: Up to approximately 30 months (through Final Analysis data cut-off of 16-May-2011)
Population: All participants who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 142
Percentage of Participants | 11.3 [6.6 to 17.7]
Statistical Analysis 1: Comparison: Vorinostat + Bortezomib; Test type: Other; p = 0.419, Exact Test for Binomial Parameter

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who experienced an AE were reported.
Time Frame: Up to approximately 22 months
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 142
Participants | 142

3. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately 18 months
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 142
Participants | 28

4. Secondary Outcome: Time To Disease Progression (TTP) as Determined by IAC Per EBMT Criteria
Description: TTP was defined as the time from allocation to the first documented disease progression (PD) as determined by IAC per EBMT criteria or death due to myeloma, whichever occurred first. PD: >25% increase in level of serum Mparaprotein, which must also be an absolute increase of at least 5g/L (500 mg/dL) and confirmed on a repeat investigation or 25% increase in 24-hour urinary light chain excretion, which must also be an absolute increase of at least 200mg/24hour and confirmed on a repeat investigation or >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10% or definitive increase in size of existing LBLs or STP or development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.8 mmol/L not attributable to any other cause). To report the median TTP (in months) and associated 95% CIs Kaplan-Meier method was used.
Time Frame: Up to approximately 30 months (through Final Analysis data cut-off of 16-May-2011)
Population: All participants who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 142
Months | 3.47 [2.53 to 4.57]

5. Secondary Outcome: TTP as Assessed by Investigator Per EBMT Criteria
Description: TTP was defined as the time from allocation to the first documented PD as assessed by investigator per EBMT criteria or death due to myeloma, whichever occurred first. PD: >25% increase in level of serum Mparaprotein, which must also be an absolute increase of at least 5g/L (500 mg/dL) and confirmed on a repeat investigation or 25% increase in 24-hour urinary light chain excretion, which must also be an absolute increase of at least 200mg/24hour and confirmed on a repeat investigation or >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10% or definitive increase in size of existing LBLs or STP or development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.8 mmol/L not attributable to any other cause). To report the median TTP (in months) and associated 95% CIs Kaplan-Meier method was used.
Time Frame: Up to approximately 30 months (through Final Analysis data cut-off of 16-May-2011)
Population: All participants who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 142
Months | 3.07 [2.37 to 4.33]

6. Secondary Outcome: Progression-Free Survival (PFS) as Determined by IAC Per EBMT Criteria
Description: PFS was defined as the time from allocation to the first documents PD as determined by IAC per EBMT criteria or death due to any cause, whichever occurs first. PD: >25% increase in level of serum M-paraprotein, which must also be an absolute increase of at least 5g/L (500 mg/dL) and confirmed on a repeat investigation or 25% increase in 24-hour urinary light chain excretion, which must also be an absolute increase of at least 200mg/24hour and confirmed on a repeat investigation or >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10% or definitive increase in size of existing LBLs or STP or development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.8 mmol/L not attributable to any other cause). To report the median PFS (in months) and associated 95%CIs Kaplan-Meier method was used.
Time Frame: Up to approximately 30 months (through Final Analysis data cut-off of 16-May-2011)
Population: All participants who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 142
Months | 3.13 [2.40 to 4.33]

7. Secondary Outcome: PFS as Assessed by Investigator Per EBMT Criteria
Description: PFS was defined as the time from allocation to the first documents PD as assessed by investigator per EBMT criteria or death due to any cause, whichever occurs first. PD: >25% increase in level of serum M-paraprotein, which must also be an absolute increase of at least 5g/L (500 mg/dL) and confirmed on a repeat investigation or 25% increase in 24-hour urinary light chain excretion, which must also be an absolute increase of at least 200mg/24hour and confirmed on a repeat investigation or >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10% or definitive increase in size of existing LBLs or STP or development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.8 mmol/L not attributable to any other cause). To report the median PFS (in months) and associated 95%CIs Kaplan-Meier method was used.
Time Frame: Up to approximately 30 months (through Final Analysis data cut-off of 16-May-2011)
Population: All participants who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 142
Months | 2.83 [2.17 to 3.77]

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from allocation to death due to any cause. To report the median survival (in months) and the associated 95%CIs were reported using Kaplan-Meier method was used. Participants without documented death at the time of final analysis were censored at the date of the last follow up.
Time Frame: Up to approximately 40 months (through End of Trial data cut-off of 09-Apr-2012)
Population: All allocated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 143
Months | 11.23 [8.47 to 14.43]

ADVERSE EVENTS:
Time Frame: Up tp approximately 22 months for non-serious adverse events (AEs). Up to approximately 40 months for serious AEs and all-cause mortality.
Description: All-Cause Mortality reported for all randomized participants. Serious AEs and Other AEs were reported for all enrolled participants who received at least 1 dose of study treatment. Only serious AEs were collected for participants treated on extension.
Arm/Group | Vorinostat + Bortezomib
All-Cause Mortality (participants affected / at risk) | 85/143
Serious Adverse Events (participants affected / at risk) | 92/142
Other Adverse Events (participants affected / at risk) | 140/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat + Bortezomib (N=142)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (8)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 6 (6)
Fatigue (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 7 (7)
Immunodeficiency (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1)
H1N1 influenza (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 13 (14)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Septic shock (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 12 (15)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30 (31)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 10 (12)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat + Bortezomib (N=142)
Anaemia (Blood and lymphatic system disorders) | 74 (231)
Leukopenia (Blood and lymphatic system disorders) | 25 (74)
Neutropenia (Blood and lymphatic system disorders) | 53 (135)
Thrombocytopenia (Blood and lymphatic system disorders) | 99 (582)
Vision blurred (Eye disorders) | 11 (13)
Abdominal discomfort (Gastrointestinal disorders) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 18 (25)
Abdominal pain upper (Gastrointestinal disorders) | 12 (18)
Constipation (Gastrointestinal disorders) | 35 (47)
Diarrhoea (Gastrointestinal disorders) | 74 (189)
Dry mouth (Gastrointestinal disorders) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 11 (16)
Nausea (Gastrointestinal disorders) | 80 (162)
Vomiting (Gastrointestinal disorders) | 53 (103)
Asthenia (General disorders) | 31 (57)
Chest pain (General disorders) | 13 (15)
Chills (General disorders) | 12 (14)
Fatigue (General disorders) | 69 (143)
Oedema peripheral (General disorders) | 17 (18)
Pyrexia (General disorders) | 34 (56)
Nasopharyngitis (Infections and infestations) | 14 (19)
Upper respiratory tract infection (Infections and infestations) | 17 (23)
Contusion (Injury, poisoning and procedural complications) | 10 (12)
Blood creatinine increased (Investigations) | 18 (31)
Platelet count decreased (Investigations) | 15 (48)
Weight decreased (Investigations) | 13 (21)
Decreased appetite (Metabolism and nutrition disorders) | 53 (78)
Dehydration (Metabolism and nutrition disorders) | 11 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (27)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (17)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (22)
Dizziness (Nervous system disorders) | 21 (26)
Headache (Nervous system disorders) | 25 (35)
Neuralgia (Nervous system disorders) | 14 (17)
Neuropathy peripheral (Nervous system disorders) | 17 (27)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (14)
Insomnia (Psychiatric disorders) | 13 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 (56)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 (36)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Haematoma (Vascular disorders) | 8 (10)
Hypertension (Vascular disorders) | 13 (17)
Hypotension (Vascular disorders) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.